CLINICAL TRIAL: NCT02929641
Title: Evaluation of a New Image-enhanced Endoscopic Technology With Magnification Using I-scan Optical Enhancement for Prediction Colorectal Polyp Histology
Brief Title: Evalution of Optical Enhancement With Magnification for Polyop Histology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Professor, Shandong University
Other Study IDs: 2016SDU-QILU-14
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Polyps
Keywords: Optical Enhancement technology; coloractal polyp prediction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HDWL and OE with magnification: The polyps found will be observed by HDWL and OE with magnicication model and recorded.

SUMMARY:
When a polyp is found, it woulf be recorded by a white-light and OE1 model with magnification for assessing and predicting its histology. After that, its really histology will be reported by an pathologist.

When a polyp is found, OE mode 1 with magnification was first used with near focus the polyp and an endoscopist made a real-time prediction of polyp pathology. After that, high-definition mode and OE mode 1 without magnification were used to observe polyp sequencely. The video of all procedure was recorded.

DETAILED DESCRIPTION:
After bowel cleansing with 2L polyethylene glycol, patients received colonoscopy under propofol intravenous anesthesia. When a polyp was found, we began to wash it and record the video. OE mode 1 with magnification was first used with near focus the polyp and an endoscopist made a real-time prediction of polyp pathology. After that, high-definition mode and OE mode 1 without magnification were used to observe polyp sequencely. Biopsy of the polyps were taken after observation, and the size of polyps was estimated by the biopsy forceps. The information of patient age, gender polyp morphology and location were recorded. After a video transcoding and clipping, the pathology type of each video clip was predicted by an endoscopist. The sensitivity, specificity, positive predicting value (PPV), negative predicting value (NPV) and accuracy were calculated. The pathology types of polyps were classified by non-neoplastic polyps and neoplastic polyps according to Vienna Classification. Statistics were performed by NCSS 11 and R software (Version 3.3.2).

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are found polyps during endoscopy procesure.

Exclusion Criteria:

* Inflammatory bowel disease
* Biopsies were not available.
* Unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who experence an examation of coloscopy found polyps.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
To evaluated the accuracy of i-scan OE system with magnification endoscopy on real-time predicting the pathology types of colorectal polyps. | 18 months
  To evaluated the accuracy of i-scan OE system with magnification endoscopy on real-time predicting the pathology types of colorectal polyps.

SECONDARY OUTCOMES:
To evaluate whether the diagnostic value of OE with magnification can meet the thresholds of "resect-and-discard" and "diagnose-and-leave" strategies outlined by Preservation and Incorporation of Valuable Endoscopic Innovations (PIVI) document. | 18 months
  To evaluate whether the diagnostic value of OE with magnification can meet the thresholds of "resect-and-discard" and "diagnose-and-leave" strategies outlined by Preservation and Incorporation of Valuable Endoscopic Innovations (PIVI) document.
To assess the diagnostic value and inter-observer agreement of OE on post-hoc differentiating pathology of colorectal polyps. | 18 months
  To assess the diagnostic value and inter-observer agreement of OE on post-hoc differentiating pathology of colorectal polyps.
To assess the value of magnification optical enhancement on classification of colorectal polyps using a deep learning model | 18 months
  To assess the value of magnification optical enhancement on classification of colorectal polyps using a deep learning model

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD,PhD, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Basford PJ, Longcroft-Wheaton G, Higgins B, Bhandari P. High-definition endoscopy with i-Scan for evaluation of small colon polyps: the HiSCOPE study. Gastrointest Endosc. 2014 Jan;79(1):111-8. doi: 10.1016/j.gie.2013.06.013. Epub 2013 Jul 17. PMID 23871094
- [Result] Neumann H, Fujishiro M, Wilcox CM, Monkemuller K. Present and future perspectives of virtual chromoendoscopy with i-scan and optical enhancement technology. Dig Endosc. 2014 Jan;26 Suppl 1:43-51. doi: 10.1111/den.12190. Epub 2013 Oct 23. PMID 24373000